CLINICAL TRIAL: NCT06760702
Title: A Phase II, Open-label, Randomized, Dose-ranging Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of AUR 109 in Patients with Colorectal, Ovarian, and Renal Cancers (TEJAS-2)
Brief Title: A Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of AUR 109 in Patients with Colorectal, Ovarian, and Renal Cancers
Acronym: TEJAS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUR109-202
Record Dates: First submitted 2024-11-07; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer; Colorectal Cancer; Renal Cancer
Keywords: Colorectal cancer; Ovarian cancer; Renal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Three Dose regimens of 200 mg, 300 mg and 400 mg with 10 patients in each dose arm, are applied to three different indications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colorectal cancer (Experimental)
  Interventions: Drug: AUR109 200mg; Drug: AUR109 300mg; Drug: AUR109 400mg
- Ovarian Cancer (Experimental)
  Interventions: Drug: AUR109 200mg; Drug: AUR109 300mg; Drug: AUR109 400mg
- Renal Cancer (Experimental)
  Interventions: Drug: AUR109 200mg; Drug: AUR109 300mg; Drug: AUR109 400mg

INTERVENTIONS:
Drug: AUR109 200mg — AUR109 200mg (once daily)
Drug: AUR109 300mg — AUR109 300mg once daily
Drug: AUR109 400mg — AUR109 400mg once daily

SUMMARY:
This is an open-label, multicentre, randomized, Phase II study and will be conducted with co-primary objectives of the study are to assess the efficacy of AUR109, as measured by ORR and safety / tolerability at three different dose levels of the study drug in three cancer indications i.e., colorectal, ovarian cancer and renal cancer.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicenter study evaluating the efficacy and safety of the drug AUR109 at three different dose levels (200 mg, 300 mg, and 400 mg) in patients with colorectal, ovarian, or renal cancer. Participants must have undergone at least two lines of systemic therapy and exhausted all local treatment options. The 200 mg and 300 mg doses will be administered continuously over a 21-day cycle, while the 400 mg dose will follow an interrupted regimen (2 weeks on, 1 week off). The drug is to be taken once daily according to the specified dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent and agree to comply with all study related activities.
* Male or female patients aged ≥ 18 years.
* Pathological diagnosis of adenocarcinoma of colorectal origin, epithelial ovarian cancer (ovarian cancer term also includes fallopian tube cancer as well as primary peritoneal cancer), or renal cell carcinoma of the kidney.
* Patients must have received at least two lines of systemic therapy and should have exhausted all available local therapies. At a minimum, for each of the respective cancer types, patients should have received the following:

Colorectal Cancer - Previous treatment should include 5-FU based treatments, oxaliplatin based treatments, irinotecan-based treatments, IV VEGF inhibitors, IV EGFR antibodies (for KRAS wildtype), PD-1 antibodies for known MSI-H positive tumors, regorafenib and lonsurf, anti-HER2 agents (e.g., FDA approved Tucatinib and Trastuzumab combination, where available) for HER2 amplified colorectal cancer, unless any of these are not available locally or prohibitive for the patient financially or if the patient is not eligible for these or if the patient has refused these.

Ovarian cancer (also includes fallopian tube cancer and primary peritoneal cancer) - Tumor must be platinum refractory, defined as treatment free interval of < 6 months from the last platinum-based regimen. In addition, patient should have received topotecan, gemcitabine, liposomal doxorubicin, bevacizumab and PARP inhibitors (for BRCA mutants), mirvetuximab for folate receptor alpha amplified ovarian cancer, unless any of these are not available locally or prohibitive for the patient financially or if the patient is not eligible for these or if the patient has refused these.

Renal Cell Carcinoma - Patient should have received an oral VEGF inhibitor and PD-1/PD-L1 inhibitors, unless any of these are not available locally or prohibitive for the patient financially or if the patient is not eligible for these or if the patient has refused these.

* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1 (Patients with disease related ECOG 2 are allowed, in addition to ECOG 0 and 1).
* Acceptable bone marrow function as described below:

ANC ≥ 1200/μL (without WBC growth factor support) Platelet count ≥ 90,000/μL without transfusion support Hemoglobin ≥ 9 g/dL (Transfusion is allowed to achieve this Hb)

* Acceptable organ function as described below:

Total Bilirubin ≤ 1.2 x ULN AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases) ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases) Creatinine clearance (CrCl) ≥ 30 mL/min (either measured or estimated by the Cockcroft- Gault formula) [Cockcroft-Gault formula for estimated creatinine clearance (eCrCl) = (140 - Age) × Weight (kg) × (0.85 if Female) / (72 × serum creatinine (mg/dL))] Albumin ≥ 3.0 g/dL

* Ability to swallow and retain oral medications.
* Negative serum pregnancy test in women of childbearing potential (WOCBP).
* Women of childbearing potential and men who partner with such a woman of childbearing potential must agree to use one or more of highly effective method(s) for contraception for the duration of the study, i.e., through 28-day follow up visit, after discontinuation of study drug(s).
* Evidence of measurable disease per RECIST, v1.1 for solid tumors. Measurable disease for solid tumors is defined as at least one lesion that can be accurately measured in at least 1 dimension with a minimum size of 10 mm for non-nodal lesions or 15 mm in short axis for nodal lesions.

Exclusion Criteria:

* Patients without any wild type allele (Such as *28/*28, *37/*37 or *37/*28 variants) genotypes for UGT1A1.
* Systemic anti-cancer therapy, such as chemotherapy, biological therapy, or Immunomodulatory drug therapy, received within the past 28 days or 5 half-lives, whichever is longer, from the Cycle 1 Day 1 of the study.
* Presence of an acute or chronic toxicity resulting from prior anti-cancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0.
* Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial).
* Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) metastases. Patients with previously treated (> 6 months of screening) and are now stable and asymptomatic, from CNS perspective, are allowed.
* Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia).
* Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness.
* Known active or chronic hepatitis B or hepatitis C infection.
* Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1.
* Left Ventricular Ejection Fraction (LVEF) < 50% at screening.
* Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1.
* The QTcF (corrected QT interval Fridericia method) value in the screening ECG > 460 ms in both males and females.
* Previous or concomitant additional malignancy, except for basal-cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix; patients with other malignancies are eligible if they have remained disease free for at least 2 years prior to trial entry and in the opinion of the investigator deemed to have a low likelihood of recurrence.
* Pregnant or lactating women.
* Any clinically significant medical, psychiatric, or social condition; or laboratory abnormality that may increase the risk of trial participation or may interfere with the informed consent process and/or with compliance with the requirements of the trial or may interfere with the interpretation of the trial results and, in the Investigator's opinion, would make the patient inappropriate for entry into this trial.
* Patients who require concomitant administration of drugs which have a high risk of prolonging QT interval.
* Availability of any therapeutic options approved locally.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 90 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy | Baseline, Cycle 2 Day 1,Cycle 4 Day 1,Cycle 6 Day1,Cycle 8 Day 1 and Cycle 10 Day 1 (each cycle is 21 days)
  To assess the safety and efficacy of three dose levels of AUR109 (200 mg, 300 mg, and 400 mg) in patients with colorectal, ovarian, and renal cancers, as measured by Objective Tumor Response Rate (ORR) (CR + PR).

SECONDARY OUTCOMES:
Pharmacokinetic Profile (Cmax) | Day 1 and Day 15
  Maximum concentration of AUR109
Pharmacokinetic Profile (Tmax) | Day 1 and Day 15
  Tmax in hours
Pharmacokinetic Profile (AUC) | Day 1 and Day 15
  Area under the curve of AUR109 in ng/ml
HRQoL | Assessment will be performed at 3 rd week (Day 15 to 21) of every 3 cycles (21 days per Cycle) until either progressive disease or intolerable toxicity occurs
  FACT-G (Functional Assessment of Cancer Therapy - General) Score (scalle range is 0 (Lowest) to 4 (Highest)

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Gindodi Devi Hospital, Khursīpār, Chhattisgarh
  - Kiran Multi Super Speciality Hospital and Research Centre, Surat, Gujarat
  - Sunshine Global Hospitals, Surat, Gujarat
  - Sujan Surgical Cancer Hospital and Amravati Cancer Foundation, Amravati, Maharashtra
  - Uro-Science Centre, S.P. Medical College & AG of Hospitals, Bikaner, Rajasthan

IPD SHARING:
Plan to Share IPD: No